CLINICAL TRIAL: NCT03672786
Title: Gene Expression in Nutritional Intervened Athletes
Brief Title: Gene Expression in Intervened Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University of La Laguna (Other)
Responsible Party: Principal Investigator, Elena Planells del Pozo, University Professor, Universidad de Granada
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI10/1993
Record Dates: First submitted 2018-09-08; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Genetic Change; Athlete
Keywords: Gene Expression; Athletes; Micronutrient Intervention; Whole Blood

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Sedentary: Multicentrum® 2 months. Subjects maintaining the multivitamin supplement (Multicentrum® (Pfizer, Spain) 1 tablet/day) during 2 months
  Interventions: Dietary Supplement: Multicentrum
- Experimental Group (Experimental): Athletes: Multicentrum® 2 months. Subjects maintaining the multivitamin supplement (Multicentrum® (Pfizer, Spain) 1 tablet/day) during 2 months
  Interventions: Dietary Supplement: Multicentrum

INTERVENTIONS:
Dietary Supplement: Multicentrum — The multivitamin supplement (Multicentrum® (Pfizer, Spain) 1 tablet/day) will be maintained during 2 months
  Other Names: Multicentrum 2 months

SUMMARY:
Background: Exercise represents an important challenge for the homeostasis of the entire body that occurs on a cellular and systemic level in which micronutrients play an important role in regulating the processes that sustain athletic performance. Objective: The investigators measured changes in gene expression of whole blood in a group of athletes and sedentary participants and compared gene modulation before and after nutritional intervention with micronutrients. Methods: Blood samples were taken from thirteen athletes and thirteen sedentary age- and gender-matched participants. The study design was carried out over a period of 4 months where three time points were established: (T0) baseline conditions in the sedentary and athlete groups; (T2) after two months of supplementation; (T4) after two months in the absence of nutritional supplementation. Differential gene expression was evaluated in 112 genes using RT-qPCR analysis with the QuantStudioTM 12K Flex Real-Time PCR System.

DETAILED DESCRIPTION:
Background: Exercise represents an important challenge for the homeostasis of the entire body that occurs on a cellular and systemic level in which micronutrients play an important role in regulating the processes that sustain athletic performance. Objective: The investigators measured changes in gene expression of whole blood in elite athletes and sedentary subjects and compared gene modulation before and after nutritional intervention with micronutrients. Methods: Thirteen elite athletes and thirteen sedentary controls were enrolled in the present study. Blood samples were taken from athletes and sedentary age- and gender-matched subjects. The study design was carried out over a period of 4 months where three time points were established: (T0) baseline conditions in the sedentary and handball groups; (T2) after two months of supplementation; (T4) after two months in the absence of nutritional supplementation. Differential gene expression was evaluated in 112 genes using RT-qPCR analysis with the QuantStudioTM 12K Flex Real-Time PCR System.

ELIGIBILITY:
Inclusion Criteria:

* To pass a recruitment medical examination consisting of a clinical examination and recording the participant's medical history.
* Non-smoker and not being on a medication regimen.
* Written informed consent prior to participation.
* With regard to the sedentary controls, none of the subjects reported at least 150 min·wk-1 of moderate-intensity or 75 min·wk-1 of vigorous-intensity aerobic physical activity necessary for substantial health benefits.
* With regard to athletes, to be involved in a training regime including both indoor exercise and integrated conditioning exercises in addition to competing in matches on weekends.

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male, Adult
Enrollment: 26 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Gene expression analysis | 6 months
  112 genes using RT-qPCR analysis with the QuantStudioTM 12K Flex Real-Time PCR System. Relative quantification was determined using the 2-ΔCT method. Cut-off punctuation was established as 1.5.

SECONDARY OUTCOMES:
Anthropometric assessment - Height | 6 months
  Anthropometric assessment recorded data were height in centimetres (SECA® Model 274).
Anthropometric assessment - Weight | 6 months
  Anthropometric assessment recorded data were weight in kilograms (Tanita MC-980 Body Composition Analyzer MA Multifrequency Segmental, Barcelona, Spain).
Anthropometric assessment - BMI | 6 months
  Anthropometric assessment recorded data BMI was calculated calculated as weight/height^2 and expressed kg/m2 equation.
Anthropometric assessment - Fat percentage | 6 months
  Anthropometric assessment recorded data BMI was measured by multifrequency bioelectrical impedance (Tanita MC-980 Body Composition Analyzer MA Multifrequency Segmental, Barcelona, Spain) and expressed in kilograms and as the percentage of body fat. Participants were informed in advance of the required conditions prior to the measurement: no alcohol less than 24 hours before the measurement, no vigorous exercise less than 12 hours prior to the measurement, no food or drink less than 3 hours prior to the measurement, and no urination immediately before the measurement. All measurements were taken simultaneously during the morning in fasting conditions.
Anthropometric assessment - Fat free mass | 6 months
  Anthropometric assessment recorded data fat free mass was measured by multifrequency bioelectrical impedance (Tanita MC-980 Body Composition Analyzer MA Multifrequency Segmental, Barcelona, Spain) and expressed in kilograms and as the percentage of fat-free mass. Participants were informed in advance of the required conditions prior to the measurement: no alcohol less than 24 hours before the measurement, no vigorous exercise less than 12 hours prior to the measurement, no food or drink less than 3 hours prior to the measurement, and no urination immediately before the measurement. All measurements were taken simultaneously during the morning in fasting conditions.
Anthropometric assessment - Muscle mass | 6 months
  Anthropometric assessment recorded data muscle mass was measured by multifrequency bioelectrical impedance (Tanita MC-980 Body Composition Analyzer MA Multifrequency Segmental, Barcelona, Spain) and expressed in kilograms. Participants were informed in advance of the required conditions prior to the measurement: no alcohol less than 24 hours before the measurement, no vigorous exercise less than 12 hours prior to the measurement, no food or drink less than 3 hours prior to the measurement, and no urination immediately before the measurement. All measurements were taken simultaneously during the morning in fasting conditions.
Biochemical parameters - Glucose | At baseline
  Biochemistry was performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®). Glucose was measured and expressed in mg/dL. The reference value is established in 70 - 110 mg/dL.
Biochemical parameters - Creatinine | At baseline
  Biochemistry was performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®). Creatinine was measured and expressed in mg/dL. The reference value is established in 0.5 - 0.9 mg/dL.
Biochemical parameters - Urea | At baseline
  Biochemistry was performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®). Urea was measured and expressed in mg/dL. The reference value is established in 10 - 50 mg/dL.
Biochemical parameters - Uric acid | At baseline
  Biochemistry was performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®). Uric acid was measured and expressed in mg/dL. The reference value is established in 2.4 - 5.7 mg/dL.
Biochemical parameters - Triglycerides | At baseline
  Biochemistry was performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®). Triglycerides acid was measured and expressed in mg/dL. The reference value is established in 50 - 200 mg/dL.
  total cholesterol (mg/dL), total proteins (g/dL), transferrin (mg/dL) and albumin (mg/dL).
Biochemical parameters - Total cholesterol | At baseline
  Biochemistry was performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®). Total cholesterol was measured and expressed in mg/dL. The reference value is established in 110 - 200 mg/dL.
Biochemical parameters - Total proteins | At baseline
  Biochemistry was performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®). Total proteins were measured and expressed in mg/dL. The reference value is established in 6.6 - 8.7 g/dL.
Biochemical parameters - Transferrin | At baseline
  Biochemistry was performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®). Transferrin was measured and expressed in mg/dL. The reference value is established in 200 - 360 mg/dL.
Biochemical parameters - Albumin | At baseline
  Biochemistry was performed after 12 hours of fasting first thing in the morning, by specialists puncturing the cubital vena cava (Venoject®). Albumin was measured and expressed in mg/dL. The reference value is established in 3.5 - 5.2 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Planells, PhD, Study Director — Universidad de Granada; Jorge Molina, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Universidad de Granada, Granada, Spain